CLINICAL TRIAL: NCT01869530
Title: TARGet Kids!: Measuring Nutrition in Young Preschool Children in the Primary Care Practice Setting
Acronym: TARGetKids!
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Catherine Birken, Staff Paediatrician, The Hospital for Sick Children
Other Study IDs: 2063
Record Dates: First submitted 2013-05-28; First posted 2013-06-05 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Nutritional Disorders; Obesity; Development
MeSH Terms: conditions — Nutrition Disorders; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy children

SUMMARY:
TARGet Kids! (The Applied Research Group for Kids) is a research study enrolling healthy children aged 0-5 years. The aim of the TARGet Kids! registry is to link early life exposures to health problems including obesity, micronutrient deficiencies, and developmental problems.

TARGet Kids! represents an innovative collaboration between child health researchers and children's primary care doctors (pediatricians and family physicians) to promote research that really matters and create solutions to some of the today's biggest health concerns. The results of this collaborative research study are not only improving the quality of children's healthcare but also the health of children across the country. Coordinated by Sick Kids and St. Michael's Hospital with data management services by the Applied Health Research Centre (AHRC), TARGet Kids! is the only primary care research network for children in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Birth to less than 6 years of age
* Parental consent
* Attending a TARGet Kids! research network practice

Exclusion Criteria:

* Chronic illness with the exception of asthma

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children are recruited from 12 pediatric and family medicine primary care practices in Toronto, Ontario, and Montreal, Quebec, Canada.
Sampling Method: Non-Probability Sample
Enrollment: 14000 (Estimated)
Dates: Start 2008-07 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | 10 years (yearly measurements)
  Change in BMI over a 10 year follow-up period

SECONDARY OUTCOMES:
Nutrition | Yearly measurements
  Nutritional risk
Development | Yearly measurements
  Child development
Mental Health | Yearly measurements
  Mental Health
Lifestyle Factors | Yearly measurements
  Assessment of Lifestyle Factors that contribute to health
Child Behavior | Yearly measurements
  Child behavior
Social Determinants | Yearly measurements
  Social determinants of health
Education | Yearly measurements
  Nutritional factors affects on education
Parenting | Yearly measurements
  Parenting styles

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - St. Michael's Hospital, Toronto, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Melville Pediatric Center, Montreal, Quebec

REFERENCES:
- [Derived] Borkhoff CM, Imsirovic H, Bayoumi I, Macarthur C, Nurse KM, To T, Feldman M, Lau E, Knight B, Birken CS, Maguire JL, Parkin PC. Developmental screening at 18 months using the Nipissing District Developmental Screen. Paediatr Child Health. 2025 May 11;30(6):477-485. doi: 10.1093/pch/pxaf023. eCollection 2025 Sep. PMID 41049705
- [Derived] Kucab MD, Keown-Stoneman CD, Birken CS, Perlman M, Parsons J, D'Annunzio D, Thadani S, Allen CA, Maguire JL; TARGet Kids! Collaboration. Center-Based Childcare in Early Childhood and Nutritional Risk in Later Childhood: A Prospective Cohort Study. J Nutr. 2025 Dec;155(12):4530-4539. doi: 10.1016/j.tjnut.2025.09.028. Epub 2025 Sep 27. PMID 41022151
- [Derived] Nurse KM, Parkin PC, Keown-Stoneman CDG, Bayoumi I, Birken CS, Maguire JL, Macarthur C, Borkhoff CM. Association Between Family Income and Positive Developmental Screening Using the Infant Toddler Checklist at the 18-Month Health Supervision Visit. J Pediatr. 2024 Jan;264:113769. doi: 10.1016/j.jpeds.2023.113769. Epub 2023 Nov 1. PMID 37821023
- [Derived] Palumbo AM, Kirkwood D, Borkhoff CM, Keown-Stoneman CDG, Muraca GM, Fuller A, Birken CS, Maguire JL, Brown HK, Anderson LN; TARGet Kids! Collaboration. Validation of Parent-reported Gestational Age Categories for Children Less Than 6 Years of Age. Epidemiology. 2023 Nov 1;34(6):767-773. doi: 10.1097/EDE.0000000000001645. Epub 2023 Sep 26. PMID 37757868
- [Derived] Braddon KE, Keown-Stoneman CD, Dennis CL, Li X, Maguire JL, O'Connor DL, Omand JA, Simpson JR, Birken CS. Maternal Preconception Body Mass Index and Early Childhood Nutritional Risk. J Nutr. 2023 Aug;153(8):2421-2431. doi: 10.1016/j.tjnut.2023.06.022. Epub 2023 Jun 24. PMID 37356500
- [Derived] Kucab MD, Keown-Stoneman CDG, Birken CS, Perlman M, Maguire JL; TARGet Kids! Collaboration. Centre-based childcare in early childhood and growth in later childhood: a prospective cohort study. Int J Obes (Lond). 2023 Aug;47(8):724-731. doi: 10.1038/s41366-023-01316-2. Epub 2023 Apr 27. PMID 37106078
- [Derived] Omand JA, Li X, Keown-Stoneman CDG, Borkhoff CM, Duku E, Lebovic G, Maguire JL, Mamdani MM, Parkin PC, Reid-Westoby C, Randall Simpson J, Tremblay MS, Janus M, Birken CS; TARGet Kids! Study Group. Body Weight at Age Four Years and Readiness to Start School: A Prospective Cohort Study. Child Obes. 2023 Jun;19(4):267-281. doi: 10.1089/chi.2022.0018. Epub 2022 Jul 13. PMID 35834646
- [Derived] Omand JA, Janus M, Maguire JL, Parkin PC, Aglipay M, Randall Simpson J, Keown-Stoneman CDG, Duku E, Reid-Westoby C, Birken CS. Nutritional Risk in Early Childhood and School Readiness. J Nutr. 2021 Dec 3;151(12):3811-3819. doi: 10.1093/jn/nxab307. PMID 34587245
- [Derived] Hamid JS, Atenafu EG, Borkhoff CM, Birken CS, Maguire JL, Bohn MK, Adeli K, Abdelhaleem M, Parkin PC. Reference intervals for hemoglobin and mean corpuscular volume in an ethnically diverse community sample of Canadian children 2 to 36 months. BMC Pediatr. 2021 May 19;21(1):241. doi: 10.1186/s12887-021-02709-w. PMID 34011305
- [Derived] Bayoumi I, Birken CS, Nurse KM, Parkin PC, Maguire JL, Macarthur C, Randall Simpson JA, Borkhoff CM. Screening for marginal food security in young children in primary care. BMC Pediatr. 2021 Apr 23;21(1):196. doi: 10.1186/s12887-021-02674-4. PMID 33892660
- [Derived] Gunaseelan V, Parkin PC, Wahi G, Birken CS, Maguire JL, Macarthur C, Borkhoff CM; Members of the TARGet Kids! Collaboration. Maternal ethnicity and iron status in early childhood in Toronto, Canada: a cross-sectional study. BMJ Paediatr Open. 2020 Apr 6;4(1):e000635. doi: 10.1136/bmjpo-2020-000635. eCollection 2020. PMID 32509978
- [Derived] Birken CS, Omand JA, Nurse KM, Borkhoff CM, Koroshegyi C, Lebovic G, Maguire JL, Mamdani M, Parkin PC, Randall Simpson J, Tremblay MS, Duku E, Reid-Westoby C, Janus M; TARGet Kids! Collaboration. Fit for School Study protocol: early child growth, health behaviours, nutrition, cardiometabolic risk and developmental determinants of a child's school readiness, a prospective cohort. BMJ Open. 2019 Nov 19;9(11):e030709. doi: 10.1136/bmjopen-2019-030709. PMID 31748293
- [Derived] Parkin PC, Koroshegyi C, Mamak E, Borkhoff CM, Birken CS, Maguire JL, Thorpe KE; TARGet Kids! Collaboration. Association between Serum Ferritin and Cognitive Function in Early Childhood. J Pediatr. 2020 Feb;217:189-191.e2. doi: 10.1016/j.jpeds.2019.09.051. Epub 2019 Nov 2. PMID 31685227
- [Derived] Wong VCH, Maguire JL, Omand JA, Dai DWH, Lebovic G, Parkin PC, O'Connor DL, Birken CS; TARGet Kids! Collaboration. A Positive Association Between Dietary Intake of Higher Cow's Milk-Fat Percentage and Non-High-Density Lipoprotein Cholesterol in Young Children. J Pediatr. 2019 Aug;211:105-111.e2. doi: 10.1016/j.jpeds.2019.03.047. Epub 2019 May 17. PMID 31104850
- [Derived] Sypes EE, Parkin PC, Birken CS, Carsley S, MacArthur C, Maguire JL, Borkhoff CM; TARGet Kids! Collaboration. Higher Body Mass Index Is Associated with Iron Deficiency in Children 1 to 3 Years of Age. J Pediatr. 2019 Apr;207:198-204.e1. doi: 10.1016/j.jpeds.2018.11.035. Epub 2019 Jan 7. PMID 30630632
- [Derived] Oatley H, Borkhoff CM, Chen S, Macarthur C, Persaud N, Birken CS, Maguire JL, Parkin PC; TARGet Kids! Collaboration. Screening for Iron Deficiency in Early Childhood Using Serum Ferritin in the Primary Care Setting. Pediatrics. 2018 Dec;142(6):e20182095. doi: 10.1542/peds.2018-2095. PMID 30487142
- [Derived] Borkhoff CM, Dai DWH, Jairam JA, Wong PD, Cox KA, Maguire JL, Birken CS, Macarthur C, Parkin PC; TARGet Kids! Collaboration. Breastfeeding to 12 mo and beyond: nutrition outcomes at 3 to 5 y of age. Am J Clin Nutr. 2018 Aug 1;108(2):354-362. doi: 10.1093/ajcn/nqy124. PMID 30101330
- [Derived] Eny KM, Chen S, Anderson LN, Chen Y, Lebovic G, Pullenayegum E, Parkin PC, Maguire JL, Birken CS; TARGet Kids! Collaboration. Breastfeeding duration, maternal body mass index, and birth weight are associated with differences in body mass index growth trajectories in early childhood. Am J Clin Nutr. 2018 Apr 1;107(4):584-592. doi: 10.1093/ajcn/nqx081. PMID 29635496
- [Derived] Anderson LN, Carsley S, Lebovic G, Borkhoff CM, Maguire JL, Parkin PC, Birken CS. Misclassification of child body mass index from cut-points defined by rounded percentiles instead of Z-scores. BMC Res Notes. 2017 Nov 28;10(1):639. doi: 10.1186/s13104-017-2983-0. PMID 29183360
- [Derived] Vanderhout SM, Birken CS, Parkin PC, Lebovic G, Chen Y, O'Connor DL, Maguire JL; TARGet Kids! Collaboration. Relation between milk-fat percentage, vitamin D, and BMI z score in early childhood. Am J Clin Nutr. 2016 Dec;104(6):1657-1664. doi: 10.3945/ajcn.116.139675. Epub 2016 Nov 16. PMID 27852618
- See also: TARGet Kids! website — http://targetkids.ca